CLINICAL TRIAL: NCT03099499
Title: A Phase 2 Study of Single Agent ONC201 in Recurrent or Metastatic Endometrial Cancer
Brief Title: Single Agent ONC201 in Recurrent or Metastatic Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Oncoceutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYN-106
Record Dates: First submitted 2017-03-23; First posted 2017-04-04 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ONC201 treatment Arm (Experimental)
  Interventions: Drug: ONC201

INTERVENTIONS:
Drug: ONC201 — ONC201 will be administered at a dose of 625 mg by mouth weekly until disease progression, unacceptable toxicity, or if the patient discontinues for any other reason. Radiologic tumor assessment would be performed at baseline, Cycle 3 Day 1, Cycle 5 Day 1, and at the end of every 3 cycles beyond cycle 5. All patients including those removed from the study due to unacceptable toxicity, will undergo radiologic tumor assessment at the time of discontinuation (End of treatment).

SUMMARY:
ONC201 is a small molecule which selectively targets the G protein-coupled receptor DRD2. Downstream of target engagement, ONC201 activates the integrated stress response (ISR) in tumor cell leading to inactivation of Akt and extracellular signal-regulated kinase (ERK) signaling as well as induction of the TRAIL pathway. ONC201 also inhibits dopamine receptor 2 (DRD2), resulting in anti-tumor responses in preclinical models. Single agent ONC201 has been examined in open-label Phase I studies in patients with advanced, treatment refractory solid malignancies. Due to its differential anti-proliferative and pro-apoptotic response in tumor cells, treatment was overall well tolerated, and the recommended phase II dose of ONC201 was set at 625mg every three weeks. An additional dose-escalation phase I study (NCT02609230) is further evaluating weekly versus three week dosing in patients with advanced solid tumors and multiple myeloma. Preliminary data from these phase I studies suggests a possible clinical benefit in patients with advanced, chemo-refractory endometrial cancers, with at least one mixed response noted in a patient with clear cell histology.

Hypothesis: Single agent ONC201 will demonstrate clinical benefit in women with recurrent or metastatic endometrial cancers, especially in those women with alterations in the Phosphoinositide 3 kinase (PI3K)/Akt/mammalian target of Rapamycin (mTOR) pathway.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed metastatic or recurrent endometrial cancer. Eligible histologies include but are not limited to endometrioid, serous, clear cell, carcinosarcoma, adenosquamous, and mixed histologies.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v. 1.1
3. Must have radiographic disease progression after 1 line of systemic cytotoxic therapy for metastatic disease or with progression within 12 months of completing adjuvant chemotherapy
4. Available archived tissue biopsies will be provided for correlative studies
5. Age > 18 years.
6. Eastern Cooperative Oncology group (ECOG) performance status of 0, 1, or 2
7. Patients must have adequate bone marrow, hepatic and renal function as defined below:

   * Leukocytes > 3,000/micro-liter (mcl)
   * Absolute neutrophil count > 1,500/mcL
   * Platelets > 100,000/mcL
   * Total bilirubin ≤1.5 upper limit of normal (ULN)
   * Aspartate aminotransferase/ Alanine aminotransferase (AST/ALT) < 2 ULN
   * Creatinine ≤1.5 ULN OR
   * Creatinine clearance > 60 Ml/min/1.73 m2 for patients with creatinine levels above ULN calculated using Calvert formula
8. Prior chemotherapy, hormonal and radiation therapy administered in the adjuvant setting will be allowed.
9. Life expectancy at least 3 months
10. Ability to understand and willingness to sign a written informed consent and HIPAA consent document
11. Patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment.

Exclusion Criteria:

1. No prior treatment with ONC201
2. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
3. The subjects who have not recovered to baseline or CTCAE ≤ Grade 1 from related toxicity to all prior therapies will be excluded. Patients with Non-serious adverse events such as alopecia, fatigue, weakness, loss of appetite and nausea that are non-significant will not be excluded.
4. Any other prior malignancy from which the patient has been disease free for less than 3 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of any site.
5. The subject is unable to swallow capsules
6. Patients receiving any other investigational agents
7. Patients with symptomatic brain metastases are excluded. Patients with asymptomatic and treated central nervous system (CNS) metastases may participate in this trial. The patient must have completed any prior treatment for CNS metastases > 28 days prior to study entry including radiotherapy or surgery. Steroids for the treatment of brain metastasis are not permitted, and patients must be stable off steroid treatment for 4 weeks prior to enrollment
8. Uncontrolled inter-current illness including, but not limited to ongoing or active infection. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism.
9. Active inflammatory gastrointestinal disease, chronic diarrhea (unless related to underlying malignancy or prior related treatment) or history of abdominal fistula, gastrointestinal perforation, peptic ulcer disease, or intra-abdominal abscess within 6 months prior to study enrollment. Gastroesophageal reflux disease under treatment with proton pump inhibitors is allowed.
10. Known Human Immunodeficiency Virus (HIV)-positive patients on combination antiretroviral therapy
11. Known history of Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection.
12. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, or in the judgment of the investigator would make the patient inappropriate for entry into the study.
13. Pregnant or breast feeding. Refer to section 4.4 for further details.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometrial cancer happens only in females
Enrollment: 19 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) rate at 12 weeks | 12 weeks
  PFS will be calculated from the day of starting the treatment until 12 weeks
Objective Response rate (ORR) as determined by Response Criteria In Solid Tumors (RECIST)1.1 criteria | 1-2 years
  ORR will be calculated from the day of starting the treatment until disease progression

SECONDARY OUTCOMES:
Safety profile of ONC201 will be determined by adverse events according to Common terminology criteria for Adverse Events (CTCAE) 4.03 | 1-2 years
  Safety profile of ONC201 will be determined by type, frequency, severity and timing and relationship of Adverse Events and lab abnormalities to ONC201
Duration of response | 1-2 years
  Duration or response will be determined from the time when a partial or complete response is seen until disease progression
Duration of stable disease | 1-2 years
  Duration of stable disease will be calculated from the time of first treatment until disease progression
Median progression free survival | 1-2 years
  Progression free survival will be calculated from the time of the start of the treatment until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Gina Mantia-Smaldone, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

FDAAA 801 VIOLATIONS:
- Violation Identified — Failure to Submit. The entry for this clinical trial was not complete at the time of submission, as required by law. This may or may not have any bearing on the accuracy of the information in the entry. — issued 2025-08-04, released 2024-12-20, posted 2025-09-03